CLINICAL TRIAL: NCT02831738
Title: Verifying Fibers Meet Regulatory Definitions for Nutrition Facts Labeling: A Randomized, Controlled Trial Evaluating Polydextrose in Dry Form
Brief Title: Fiber Effects on Glycemic Index
Acronym: PDX2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB2016-054
Record Dates: First submitted 2016-07-11; First posted 2016-07-13 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Healthy
Keywords: Fiber; Polydextrose; Glycemic Index
MeSH Terms: interventions — polydextrose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Treatment (Experimental): Polydextrose 12 g
  Interventions: Dietary Supplement: Polydextrose
- Control Treatment (Placebo Comparator): No polydextrose
  Interventions: Dietary Supplement: Control Treatment

INTERVENTIONS:
Dietary Supplement: Polydextrose — Polydextrose 12 g
  Arms: Active Treatment
Dietary Supplement: Control Treatment — no polydextrose
  Arms: Control Treatment

SUMMARY:
Primary outcome measure: Changes in plasma glucose concentration over a 3 hour postprandial visit after administration of polydextrose (12g) compared to 0 mg placebo.

Secondary outcome measure: Changes in gastrointestinal tolerance and acute bowel changes in 3 days following treatment administration.

DETAILED DESCRIPTION:
This study is a randomized, 2-arm, single-blinded, controlled, cross-over trial design focused on determining the health benefits associated with Polydextrose intake.

A planned sample size of 20 will be enrolled into the study. This study will require one initial screening visit and 2 weekly study visits. This study will take approximately 2-3 weeks per subject to complete both 3-hr study visits on two different occasions.

The initial screening visit will provide subject with the informed consent document and determine subject eligibility through anthropometric measurements, vital signs, fasting blood glucose test (finger prick), and completion of a survey relate to general eating, health, and exercise habits.

If willing and eligible to participate, subjects will be invited to participate in the study for 2 study visits. Subjects will be instructed to maintain their usual diet pattern and physical activity throughout study duration. A dinner meal will be provided the day before the study visit to control the second meal effect from the food and beverage intake of the night before the study visit.

Subject will arrive at the center in a fasted state for at least 10 hours, well hydrated and rested. Each study visit will require blood draws throughout the visit. After evaluation of subject's health status (via anthropometric, vital sign and blood glucose measurements and in-person interview), a Licensed health Care Professional will place a catheter in subject's arm for the purpose of multiple blood sample collections and take the initial blood draw in the fasting state. Subjects will be randomized to receive a placebo or test food based on randomized treatment sequences for 2 study visits on two different occasions. The sequences of receiving the test food at each visit will be randomly assigned to one of sequences.

Each study visit will involve with blood samples collection at time points 0 (fasting), 0.5, 1, 2, 3 hour (h) for assessment of change in plasma glucose concentrations.

ELIGIBILITY:
Inclusion Criteria:

* *Subject is male or female aged between 20 and 55 years of age

  * Subject has BMI between 20.0 and 32.0 kg/m2 at the screening visit
  * Fasting blood sugar less than 126 mg/dL
  * Subject is willing to maintain a stable body weight and to follow his/her regular diet and physical activity patterns throughout the study period.
  * Subject is willing to refrain from vigorous physical activity and consumption of alcoholic and/or caffeinated beverages 24 h prior to each test day
  * Subject does not smoke or has abstained from smoking for at least 2 years
  * No clinical evidence of cardiovascular, metabolic, respiratory, renal, gastrointestinal or hepatic disease
  * Not taking any medications or dietary supplements that would interfere with outcomes of the study.
  * Subject typically consumes a low fiber diet that correlates with the average fiber intake of typical western diet.

Exclusion Criteria:

* *Subject currently smokes or has smoked within the past 2 years

  * Men and women with known or suspected food intolerance, allergies or hypersensitivity to the study materials or closely related compounds
  * Men and women known to have/diagnosed with diabetes mellitus
  * Men and women with a fasting blood glucose concentration ≥126 mg/dL
  * Average blood pressure > 140 mmHg/90 mmHg during screening visit
  * Men and women with documented vascular disease, e.g., heart failure, myocardial infarction, stroke, angina, related surgeries
  * Men and women with cancer other than non-melanoma skin cancer in previous 5 years
  * Men and women who are taking medication or dietary supplements that may interfere with the outcomes of the study. Subjects may choose to go off dietary supplements (requires 30 days washout)

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-07-02 (Actual); Primary Completion 2016-08-30 (Actual); Study Completion 2016-10-25 (Actual)

PRIMARY OUTCOMES:
Changes in plasma glucose concentration over a 3 hour Postprandial Test day after administration of Polydextrose (12g) compared to Placebo (0 g) | 3 hours
  plasma glucose concentration over a 3 hour Postprandial Test day

SECONDARY OUTCOMES:
Changes in gastrointestinal tolerance using the questionnaire in 3 days following treatment administrations. | 3 days
  Gastrointestinal tolerance using the questionnaire in 3 days following treatment administration

CONTACTS AND LOCATIONS:
Overall Officials: Britt M Burton-Freeman, Ph.D, Principal Investigator — Illinois Institute of Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No